CLINICAL TRIAL: NCT05245578
Title: Skin Irritation and Phototoxicity Study of KX01 Ointment 1% in Japanese Healthy Male Subjects
Brief Title: Safety Evaluation of KX01 Ointment 1% in Japanese Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PharmaEssentia (Industry)
Collaborators: PharmaEssentia Japan K.K. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B21-101
Record Dates: First submitted 2021-12-30; First posted 2022-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Healthy Volunteer
Keywords: Skin Irritation; Phototoxicity
MeSH Terms: conditions — Dermatitis, Phototoxic

STUDY DESIGN:
Masking Description: Masking: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- KX01 ointment and Placebo ointment (Experimental)
  Interventions: Drug: KX01 ointment 1%; Drug: Placebo ointment

INTERVENTIONS:
Drug: KX01 ointment 1% — A total of 4 application sites (2 cm x 2 cm each) will be marked on each subject's back, placing 2 sites for KX01 ointment 1% and 2 sites for Placebo ointment. One set (KX01 ointment 1% and Placebo ointment patches) will be designated for irradiation and the other set will remain non-irradiated under open conditions.
Drug: Placebo ointment — A total of 4 application sites (2 cm x 2 cm each) will be marked on each subject's back, placing 2 sites for KX01 ointment 1% and 2 sites for Placebo ointment. One set (KX01 ointment 1% and Placebo ointment patches) will be designated for irradiation and the other set will remain non-irradiated under open conditions.

SUMMARY:
Skin Irritation and Phototoxicity Study of KX01 Ointment 1% in Japanese healthy male subjects

DETAILED DESCRIPTION:
A baseline evaluation of the patch sites will be performed immediately prior to application of the patches to ensure that no conditions, markings, or coloration of the skin will interfere with interpretation of the study results.

A total of 4 application sites (2 cm x 2 cm each) will be marked on each subject's back, placing 2 sites for KX01KX2-391 ointment 1% and 2 sites for Placebo vehicle ointment. One set (KX01 ointment 1% IP and Placebo ointment vehicle patches) will be designated for irradiation and the other set will remain non-irradiated under open conditions. The distance between the patches will be no less than one centimeter.

The numbering of the test sites will remain the same throughout the study. The sites will be marked with an indelible, surgical marker.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese male adult, whose age 20-65 years old

Exclusion Criteria:

* History of photosensitivity or photoallergy

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2021-11-22 (Actual); Study Completion 2022-01-12 (Actual)

PRIMARY OUTCOMES:
Degree of skin irritation at application site | 9 days
  Degree of skin irritation will be evaluated according to the criteria (response scores and response notations). The same evaluator, if possible, should perform the assessment throughout the study.
Phototoxic potential at application site | 9 days
  Phototoxic potential will be evaluated according to the criteria (response scores and response notations). The same evaluator, if possible, should perform the assessment throughout the study.

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety | 9 days

CONTACTS AND LOCATIONS:
Overall Officials: Hisakuni Sekino, Principal Investigator — Medical Corporation HOUEIKAI, Sekino Clinical Pharmacology Clinic
Locations (1):
- Medical Corporation HOUEIKAI, Sekino Clinical Pharmacology Clinic, Toshima-ku, Tokyo, Japan